CLINICAL TRIAL: NCT06264947
Title: Efficacy of Laser Acupuncture on Zanzhu (BL02) as the Treatment for Dry Age-related Macular Degeneration: A Randomized Controlled Trial
Brief Title: Efficacy of Laser Acupuncture on Zanzhu (BL02) for Dry Age-related Macular Degeneration
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Yu-Chen Lee, director of department of acupuncture, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMUH112-REC2-141
Record Dates: First submitted 2024-02-06; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Age-related Macular Degeneration
Keywords: Laser Acupuncture; Acupuncture; Age-related Macular Degeneration; Randomized Controlled Trials
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laser acupuncture group (Experimental): 3 minutes for each time, and 3 times per week, with duration of 4 weeks
  Interventions: Device: laser acupuncture
- sham laser acupuncture group (Sham Comparator): 3 minutes for each time, and 3 times per week, with duration of 4 weeks
  Interventions: Device: sham laser acupuncture

INTERVENTIONS:
Device: laser acupuncture — wavelength: 808nm energy: 18j power: 100mw
  Arms: laser acupuncture group
Device: sham laser acupuncture — wavelength: 0nm energy: 0j power: 0mw
  Arms: sham laser acupuncture group

SUMMARY:
This study is to see if laser acupuncture is a better way to treat dry-AMD (Age-related Macular Degeneration) compared to sham laser acupuncture, in the aspect of visual acuity. Investigators planed to recruit participants who are diagnosed with dry-AMD, and not younger than 20 years old. Before the study, investigators will measure the participants' BCVA (Best Corrected Visual Acuity), and then practice laser acupuncture and sham-laser acupuncture on experiment group and control group respectively. After the 4-week study, investigators will measure the participants' BCVA again.

DETAILED DESCRIPTION:
This study consists of 15 visits, which are divided into the screening period and the treatment period.

Screening visit After being provided with sufficient information for this study, the patient would voluntarily sign the informed consent. The patients who have submitted the informed consent will undergo screening tests to determine their eligibility. The screening tests include general medical history taking, treatment history for AMD, vision test. Based on the eligibility criteria and screening tests, identification codes would be granted to eligible participants.

Visit 1 Visit 1 will be arranged within a week from the screening visit. The participants who have successfully completed the screening visit can proceed to visit 1 on the same day. The participant's changes in medical history and medication taking since the screening visit will be surveyed. Randomization will be performed on the eligible participants. Before implementing each intervention, examinations would be conducted to measure outcomes, BCVA. The participants would be educated according to the assigned intervention. The experimental group would receive laser acupuncture treatment, and the control group would receive the sham laser acupuncture. In both group, any discomfort or adverse events (AEs) before and after the treatment would be surveyed. Some observation items, including vital signs, vision test, medical history, medication taking, participant's compliance, discomfort before and after the treatment and AEs, will be examined every visit. Participant teaching would also be conducted during every visit.

Visits 2-12 During visits 2-12, the observation items will be examined including visual acuity, medical history, medication taking, discomfort before and after the treatment and AEs since the last visit. Both group would visit three times a week for 4 weeks. At each visit, the experimental group would receive the laser acupuncture treatment, and the control group would receive the sham laser acupuncture. In both group, discomfort before and after the treatment would be surveyed.

Visit 13 Visit 13 will be arranged within 3 days, after a 4-week period has elapsed since visit 1. (If 4 hours have elapsed since the treatment of visit 12, visit 13 could be arranged on the same day as visit 12.) For both group, a survey would be conducted to check any changes related to medical history, medication taking and AEs since visit 12. Vision test will be conducted. When the assessments have finished, treatment satisfaction will be evaluated.

Visit 14 Visit 14 will be arranged within 3 days, after a 6-week period has elapsed since visit 1. Any changes in medical history, medication taking and AEs since visit 13 will be surveyed. Final assessments for vision test will be conducted. Lastly, the participants' final compliance will be investigated.

Additional visits Additional visits can be arranged on the participants' request or if the investigators deem them necessary. Additional follow-ups for the appeared AEs could also be arranged. They would be permitted if the AEs continue until the trial is fully completed or stopped early, or if the investigators or the participants request additional follow-ups after finishing the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Those who have been diagnosed with dry-AMD
2. Male or female patients above 20 years of age at the screening visit
3. Those who voluntarily signed the informed consent

Exclusion Criteria:

1. Those who refuse to sign the consent form
2. Pregnant women
3. Individuals with epilepsy
4. Patients with angina
5. Individuals with hyperthyroidism
6. Patients with a cardiac pacemaker
7. Those who applied immunosuppressive agents containing Arsenic

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
BCVA (Best Corrected Visual Acuity) | "baseline (pre-intervention)", and "immediately after the intervention"
  BCVA is the best possible vision an eye can see with corrective lenses. The gold standard for measuring BCVA is with the Early Treatment Diabetic Retinopathy (ETDRS) chart. The ETDRS score is calculated as the total number of letters correctly read at 4m from the chart plus 30 (if 20 or more letters can be read at 4m). If fewer than 20 letters can be read at 4m, the patient's position is adjusted to 1m in front of the chart.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chen Lee, M.D. & Ph.D., Study Director — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan